CLINICAL TRIAL: NCT04330118
Title: Origin and Function of Eosinophilic Polynuclear During Drug Reaction With Eosinophilia and Systemic Symptoms (DRESS) Syndrome
Brief Title: Origin and Function of Eosinophilic Polynuclear During DRESS Syndrome
Acronym: DRESSEO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Société de Dermatologie Française (Other); Société de Recherche en Dermatologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019_01; 2019-A02026-51 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Drug Hypersensitivity; DRESS Syndrome
Keywords: DRESS syndrome; Drug hypersensitivity; eosinophils; allergy
MeSH Terms: conditions — Drug Hypersensitivity; Drug Hypersensitivity Syndrome; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood sample
  * Serum
  * peripheral blood mononuclear cell
  * skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 20 patients with DRESS syndrome
- 20 patients with drug induced MPE with eosinophilia: patients with drug induced maculopapular exanthema (MPE) with eosinophilia
- 20 patients with drug induced MPE without eosinophilia
- 20 Healthy subjects

SUMMARY:
Drug Hypersensitivity Syndrome or DRESS for "Drug Reaction with Eosinophilia and Systemic Symptoms" is a serious drug allergy which can be life-threatening for patients with serious organ damage. The pathophysiology of DRESS is still not fully understood. In particular, no study has focused on the characterization of eosinophils, while paradoxically eosinophilia is one of the diagnostic criteria. Likewise, there is no data about the origin of eosinophils and few data are available concerning immune polarization of T-cells or the involvement of innate lymphoid cells type 2 in the recruitment of eosinophils. Our preliminary data on increase activation markers membrane expression of cutaneous eosinophils suggest that this approach could allow the identification of endotypes in which eosinophils are involved and contribute to organ damages. The correlation between tissue infiltration of eosinophils and their degree of activation would then justify the development of targeted therapeutic strategies in DRESS syndrome (anti-IL-5 therapy?). The aim of the project is: 1) Evaluate the activation status of circulating and cutaneous eosinophils in patients with DRESS compared with drug induced maculopapular exanthema without or with eosinophilia (but do not fulfill DRESS criteria) and healthy subjects; 2) Understand the pathophysiological mechanisms at the origin of this eosinophilia.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (DRESS): adult with a diagnosis of DRESS based on the following four criteria:

* Cutaneous rash occurring at least 24 hours and at most 2 months after continuous medication use
* Fever over 38 degre celcius
* At least one organ dysfunction among:
* Lymphadenopathy
* hepatitis
* Pulmonary involvement
* Cardiac involvement: myocarditis, pericarditis
* Renal impairment
* At least one of the following hematological anomalies:
* Eosinophilia ≥ 500 / mm3 .
* RegiSCAR Score ≥ 4

Groups 2 and 3 (Drug induced maculopapular exanthema without or with eosinophilia).

* Adult with drug-induced rash
* Without clinical criteria of severity defined by Djien among :
* An evolution of more than 21 days
* with organ damage as defined in group 1

Group 2 (MPE without eosinophilia): blood eosinophils < 500 / mm3

Group 3 (MPE with eosinophilia): blood eosinophils ≥ 500 / mm3

Exclusion Criteria:

* Other cause of eosinophilia including cancer, blood disease before the introduction of suspected molecule(s).
* On going oral or local corticosteroid therapy, anti-leukotriene therapy (MONTELUKAST) by the month preceding the study;
* Anti-IgE therapy (OMALIZUMAB, LIGELIZUMAB), anti-IL-5 therapy (MEPOLIZUMAB, BENRALIZUMAB) or anti-IL4 and / or anti-IL13 therapy (DUPILUMAB, TRALOKINUMAB) in the 6 months preceding the study.
* Any pregnant or lactating woman.
* Contraindication related to the blood volume taken for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with drug induced rash (DRESS, maculopapular exanthema) and healthy patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Activation status of circulating eosinophils by flow cytometry | Baseline

SECONDARY OUTCOMES:
Mean fluorescence intensity of CCR3 and IL-5R markers | Baseline
Percentage of Th2 polarized T cells | Baseline
Percentage of ILC2 | Baseline
Serum levels (ELISA) of inflammatory markers | Baseline
Correlation between the number of activated circulating eosinophils, area degranulation and severity of DRESS | Baseline
Density of extracellular granules (degranulation area and number / mm2) on skin biopsies | Baseline
NGS analysis of rearrangements of TCR (T cell receptor) | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Staumont-Salle, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (11):
- France (11):
  - CH d'Arras, Arras
  - CH de Boulogne, Boulogne-sur-Mer
  - Assistance Publique - Hôpitaux de Paris - HENRI MONDOR, Créteil
  - CH de Douai, Douai
  - CH de Dunkerque, Dunkirk
  - CH LENS, Lens
  - Hop Claude Huriez Chr Lille, Lille
  - Groupe Hospitalier de l'Institut Catholique de Lille, Lille
  - CH de Roubaix, Roubaix
  - Hôpital FOCH, Suresnes
  - CH de Valenciennes, Valenciennes